CLINICAL TRIAL: NCT06822478
Title: Randomized Blinded Clinical Trial to Evaluate the Safety and Efficacy of Arnica Tincture in the Topical Treatment of Cutaneous Leishmaniasis.
Brief Title: Arnica Tincture Fot the Treatment of Cutaneous Leishmaniasis II.
Acronym: ARNICA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: INNOVATION CORPORATION FOR THE DEVELOPMENT OF PRODUCTS FOR TROPICAL DISEASES (CIDEPRO) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEC01_2025
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Leishmaniasis, Cutaneous
Keywords: Leishmaniasis; Cutáneo; Tintura de árnica
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis | interventions — Arnicae flos extract; Solutions; Meglumine Antimoniate

STUDY DESIGN:
Intervention Model Description: This is a single-center, single-blind, randomized, comparative study with two arms. After the informed consent process and verification of the eligibility criteria, volunteers will be randomly assigned to one of the interventions: 1: Arnica tincture, topical, with 3 applications per day for 30 days; 2: intralesional pentavalent antimonials for 5 weeks (1 application per week at a dose according to the lesion area).
  After initiation of treatment, a mid-treatment telephone or face-to-face follow-up will be performed depending on the treatment arm, in addition, follow-up visits will be made at the end of treatment (+ 7 days), day 45 post-treatment (+ 5 days) and day 90 post-treatment (+ 15 days) with an optional visit on day 105 post-treatment (+ 10 days), to evaluate the response to treatment and the safety of the treatment. The participant will keep a record of study medication application to document compliance with treatment and any symptoms experienced during treatment.
Who Masked: Investigator
Masking Description: The study was designed with a single-blind design where the investigator, who performs the role of efficacy evaluator, is unaware of the treatment arm to which the participant was assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regime 1. arnica tincture (Experimental): Regimen 1: tincture of arnica applied 3 times a day for 30 days. The participant applies the tincture in the morning, afternoon and evening, that is, three times a day.
  Interventions: Drug: Arnica Tincture
- Regime 2 Pentavalent antimonials intralesionally. (Active Comparator): Administered intralesionally. At a dose of 0.008 ml X mm of area of each lesion, maximum 15 ml in total, once a week for 5 weeks.
  Interventions: Drug: Meglumine antimoniate.

INTERVENTIONS:
Drug: Arnica Tincture — Arnika tincture is a topical plant-based preparation legally authorized in Colombia and in the countries of the European community, the product of this study is Arnika tinktur Gehrlicher (5249), manufactured by Gehrlicher Pharmazeutische Extrakte GmbH, Germany. According to the European Pharmacopoeia, the solution is a 70% hydroethanolic tincture prepared from the flowers of A. montana L, and composed at least 0.04% of sesquiterpene lactones. Arnica tincture will be applied topically by each participant on all lesions until day 30.
  Other Names: topical solution
  Arms: Regime 1. arnica tincture
Drug: Meglumine antimoniate. — Monotherapy with intralesional pentavalent antimonials is one of the treatments of care used for LC in Colombia and will be used as a comparator for safety evaluation.
  Pentavalent antimonials: administered intralesionally. At a dose of 0.008 ml X mm of area of each lesion, maximum 15 ml in total, once a week for 5 weeks.
  Other Names: intralesionally; Pentavalent antimonials
  Arms: Regime 2 Pentavalent antimonials intralesionally.

SUMMARY:
Cutaneous leishmaniasis (CL) is a parasitic disease caused by more than 20 different species of the protozoan parasite Leishmania. CL usually begins with a papule at the site of the sandfly bite, which enlarges to form a nodule that progresses to an ulceration, or a scaly or warty plaque, over a period of 1 to 3 months.

The exact incidence of CL is not known. An estimated 1.2 million cases/year in approximately 100 countries worldwide suffer from different forms of CL. More than 90% of CL cases occur in the Americas and Eastern Mediterranean regions. Afghanistan, Algeria, Brazil, Colombia, Iraq, Pakistan, and Syria report more than 80% of new CL cases worldwide. Since 2010, the World Health Organization has insisted on the need to work on products that become alternatives for the treatment of LC, especially in products that can be applied topically because with them the probability of systemic toxicity is lower, increasing patient safety.

Currently, it is recommended to apply local treatments for patients with localized LC, either with pentavalent antimonials administered intralesionally or with thermotherapy. Among the options for topical treatment are natural products that have been, are and will be of utmost importance as sources of medicinal agents. In addition to natural products that have found direct medicinal applications as pharmaceutical entities, many others can serve as chemical models or templates for the design, synthesis and semi-synthesis of novel substances for the treatment of human diseases.

Arnica montana L. is a plant with anti-emollient, healing, anti-inflammatory, analgesic and antineuralgic properties; it is included in the Colombian vademecum of medicinal plants.

In a randomized phase Ib/II clinical trial conducted in patients with localized LC in Colombia, 100% (per protocol analysis) and 92% (intention-to-treat analysis) efficacy was demonstrated, with no adverse effects other than those expected such as erythema, burning, pain or itching.

By demonstrating that arnica tincture is effective and safe, and that A. montana flower extracts in different preparations (topical solutions, tinctures, liniments, ointments or gels) are approved by the European Medicines Agency and are included in the vademecum of Colombian plants issued by the Ministry of Social Protection of Colombia in 2008, the present study aims to establish the safety and efficacy of arnica tincture as an alternative for the topical treatment of localized LC compared to a currently available local therapeutic alternative: intralesional pentavalent antimonials.

DETAILED DESCRIPTION:
The exact incidence of LC is not known. For nearly 80 years, pentavalent antimony compounds: sodium stibogluconate (Pentostan®, produced by Glaxo-Wellcome) and meglumine antimoniate (Glucantime®, produced by Sanofi-Aventis) have been considered the first choice treatments for this disease despite their toxicity, difficult administration and high cost. A dose of 20 mg Sb5/kg/day for 20 days administered intramuscularly or parenterally is recommended in adult patients diagnosed with LC caused by L. braziliensis, L. panamensis, L. amazonensis, L. peruviana or L. mexicana. Pentavalent antimonials have many disadvantages such as parenteral administration and reversible side effects such as nausea, vomiting, muscle and abdominal pain, cardiac problems, increased hepatic aminotransferase concentration and chemical pancreatitis. In addition, adherence to treatment is affected by its duration (several weeks) and its availability due to restrictions on its distribution.

Since 2005, Miltefosine (hexadecylphosphocholine), an oral drug, has been proposed as the drug of first choice, especially in children diagnosed with LC caused by L. panamensis, L. mexicana, L. guyanensis or L. braziliensis; however, because it is potentially teratogenic, it is contraindicated during pregnancy and requires appropriate counseling of female patients of childbearing age and their partners in order to avoid pregnancies up to two months after the end of treatment. A dose of 50 mg for 28 days is recommended.

It is currently recommended to apply local treatments for patients with localized LC, either with pentavalent antimonials administered intralesionally or with thermotherapy. It is important to note that it is not mandatory to identify the Leishmania species to initiate treatment; however, if the most prevalent species in the region is known, treatment should be initiated according to the clinical condition of the patient, the availability of the drug and the risk-benefit balance.

PAHO recommends the use of local treatments for LC in situations in which the patient presents between 1 to 3 lesions, located in any area (except the head and periarticular areas), each lesion with an area of up to 900 mm2, with the absence of immunosuppression and the possibility of follow-up.

Arnica montana L. is a plant belonging to the Asteraceae family, which is composed of 28 to 32 species. This plant is endemic to central and southern Europe (Pyrenees and Alps), southern Scandinavia and northern Spain. It is a medicinal plant of ancestral use, recognized by several countries to alleviate various ailments. Its variety of indications can be explained by the production of a large amount of secondary metabolites such as sesquiterpene lactones (LST), flavonoids or phenolic acids. It has been demonstrated that arnica LSTs permeate through porcine skin and human skin, most of them (97%) are absorbed after 48 h and are retained in the skin, binding irreversibly to skin proteins, accumulating in the epidermis; suggesting that they do not reach systemic circulation being a safer and more beneficial treatment at local level.

The main indication corresponds to its anti-inflammatory activity. Helenalin-like LST (HL) and 11-α-13 dihydrohelenalin (DHL) are the constituents responsible for this effect, since these molecules decrease inflammation mediated by the transcription factor NF-kB. Additionally, there are other properties demonstrated in the literature such as antioxidant, antimicrobial or insecticidal activities.

Arnica tincture is a topical preparation based on the plant legally authorized in the countries of the European community and is included in the vademecun of medicinal plants in Colombia. The product under investigation is the commercial phytotherapeutic product Arnica Tintura Gehrlicher 100 mL manufactured by Gehrlicher Pharmazeutische Extrakte GmbH. According to the European Pharmacopoeia, the solution is a 70% hydroethanolic tincture prepared from the flowers of Arnica montana L., and compounded with at least 0.04% sesquiterpene lactones.

A randomized phase Ib/II clinical trial conducted in patients with localized LC in Colombia showed an efficacy of 100% (per protocol analysis) and 92% (intention-to-treat analysis), with no adverse effects other than those expected such as erythema, burning, pain or pruritus.

1. Main objectives

   * To evaluate the safety of arnica tincture in individuals with localized LC, by measuring occurrence and severity analysis of Adverse Effects (AEs), compared to treatment with pentavalent antimonials administered intralesionally.
   * To evaluate the efficacy of arnica tincture in individuals with localized LC, according to the percentage of individuals and number of lesions with clinical healing corresponding to day 90 post-treatment, compared to treatment with pentavalent antimonials administered intralesionally.
2. Secondary objectives.

   * To evaluate the frequency and severity of AEs associated with the use of arnica tincture compared to treatment with intralesionally administered pentavalent antimonials.
   * To evaluate the status of lesions over time to evidence of complete epithelialization/flattening of lesions, proportion of individuals with 100% epithelialization/flattening of lesions, and the number of epithelialized/non-indurated lesions in patients treated with tincture of arnica compared to treatment with intralesionally administered pentavalent antimonials.
   * To compare the safety and efficacy of arnica tincture with treatment with intralesionally administered pentavalent antimonials.

To evaluate the overall risks and benefits of treatment with arnica tincture compared to treatment with intralesionally administered pentavalent antimonials.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet the following inclusion criteria may enter the study and receive arnica tincture or intralesional pentavalent antimonials:

1. Males or females, over 12 years of age and adults without age limit. With a confirmed parasitological diagnosis of a primary infection of LC in at least one lesion, made by one of the following methods: 1) microscopic identification of amastigotes in the lesion tissue; 2) diagnosis of leishmania by PCR; 3) positive culture for promastigotes (Annex 2).

3. With clinical diagnosis of localized LC. 4. Ulcer, nodule or plaque type lesions. Up to 9 lesions in total, and that the total area of all lesions is ≤1875 mm2 6. Subjects who have given written IC/Assent. 7. Subject is able to understand and comply with the requirements of the study. 8. Subjects who are able to attend the control visits.

Exclusion Criteria:

Participants presenting one or more of the following criteria should be excluded from the study:

1. Diagnosis or suspicion of mucosal/mucocutaneous, diffuse or disseminated Leishmaniasis or relapse or reactivation of an LC.
2. Subjects with lesions involving the auricular region, orbital region, nasal region and/or labial region of the face, joints or in places that, in the opinion of the investigator, are difficult to apply topically or intralesionally to the study medication.
3. History of clinically significant cardiovascular, renal, hepatic, hepatic, neurological or immunological diseases that may interact positively or negatively with the treatment.
4. Having received treatment for Leishmaniasis or other treatment that, in the judgment of the investigator, may modify the course of infection with Leishmania in the last 8 weeks (56 days) prior to admission.
5. Women with a positive pregnancy test during the screening process, or lactating, or women of childbearing age who do not agree to the use of contraceptives during treatment and until DPT45.
6. Known or suspected history of hypersensitivity or idiosyncratic reactions to the investigational product or pentavalent antimonials in the trial.
7. Subjects who are unwilling to attend study visits or who are unable to comply with follow-up visits for up to three months.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with healing (scarring) after treatment | day 90
  Defined as 100% epithelialization of the lesion (s) by day 90 post-treatment.

SECONDARY OUTCOMES:
Number of participants with Final post-treatment Healing | day 105
  initial cure with no recurrence and/or mucosal involvement at 90 days post-treatment evaluation to 105 days.
  If the subject is withdrawn from the study because the lesion(s) are not healing, then the subject will also be considered a treatment failure. Any subject who has not had the lesion assessed at the scheduled times up to DPT105 will also be considered a failure in the ITT analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Iván D Velez, PhD, Principal Investigator — Clinical research group -Program for Research and Control in Tropical Diseases GIC - PECET, Medellín, Antioquia
Locations (1):
- Grupo de Investigación Clínica PECET (GIC-PECET), Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jurgens FM, Herrmann FC, Robledo SM, Schmidt TJ. Dermal Absorption of Sesquiterpene Lactones from Arnica Tincture. Pharmaceutics. 2022 Mar 29;14(4):742. doi: 10.3390/pharmaceutics14040742. PMID 35456576
- [Background] Guidelines of the International Conference on Harmonization - Good Clinical Practice: Consolidated Guide (ICH E6), E6(R2) Current Step 4 version dated 9 November 2016
- [Background] Iannitti T, Morales-Medina JC, Bellavite P, Rottigni V, Palmieri B. Effectiveness and Safety of Arnica montana in Post-Surgical Setting, Pain and Inflammation. Am J Ther. 2016 Jan-Feb;23(1):e184-97. doi: 10.1097/MJT.0000000000000036. PMID 25171757
- [Background] Wagner S, Suter A, Merfort I. Skin penetration studies of Arnica preparations and of their sesquiterpene lactones. Planta Med. 2004 Oct;70(10):897-903. doi: 10.1055/s-2004-832613. PMID 15490315
- [Background] Velasco-Castrejon O, Walton BC, Rivas-Sanchez B, Garcia MF, Lazaro GJ, Hobart O, Roldan S, Floriani-Verdugo J, Munguia-Saldana A, Berzaluce R. Treatment of cutaneous leishmaniasis with localized current field (radio frequency) in Tabasco, Mexico. Am J Trop Med Hyg. 1997 Sep;57(3):309-12. doi: 10.4269/ajtmh.1997.57.309. PMID 9311641
- [Background] Lopez L, Robayo M, Vargas M, Velez ID. Thermotherapy. An alternative for the treatment of American cutaneous leishmaniasis. Trials. 2012 May 17;13:58. doi: 10.1186/1745-6215-13-58. PMID 22594858
- [Background] Lee SA, Hasbun R. Therapy of cutaneous leishmaniasis. Int J Infect Dis. 2003 Jun;7(2):86-93. doi: 10.1016/s1201-9712(03)90002-6. PMID 12839708
- [Background] Reveiz L, Maia-Elkhoury AN, Nicholls RS, Romero GA, Yadon ZE. Interventions for American cutaneous and mucocutaneous leishmaniasis: a systematic review update. PLoS One. 2013 Apr 29;8(4):e61843. doi: 10.1371/journal.pone.0061843. Print 2013. PMID 23637917
- [Background] Alvar J, Velez ID, Bern C, Herrero M, Desjeux P, Cano J, Jannin J, den Boer M; WHO Leishmaniasis Control Team. Leishmaniasis worldwide and global estimates of its incidence. PLoS One. 2012;7(5):e35671. doi: 10.1371/journal.pone.0035671. Epub 2012 May 31. PMID 22693548
- [Background] Votypka J, Kasap OE, Volf P, Kodym P, Alten B. Risk factors for cutaneous leishmaniasis in Cukurova region, Turkey. Trans R Soc Trop Med Hyg. 2012 Mar;106(3):186-90. doi: 10.1016/j.trstmh.2011.12.004. Epub 2012 Jan 26. PMID 22284721
- [Background] Croft SL, Seifert K, Yardley V. Current scenario of drug development for leishmaniasis. Indian J Med Res. 2006 Mar;123(3):399-410. PMID 16778319
- [Background] Velez I, Lopez L, Sanchez X, Mestra L, Rojas C, Rodriguez E. Efficacy of miltefosine for the treatment of American cutaneous leishmaniasis. Am J Trop Med Hyg. 2010 Aug;83(2):351-6. doi: 10.4269/ajtmh.2010.10-0060. PMID 20682881
- [Background] Herwaldt BL. Leishmaniasis. Lancet. 1999 Oct 2;354(9185):1191-9. doi: 10.1016/S0140-6736(98)10178-2. PMID 10513726
- [Background] Tiuman TS, Santos AO, Ueda-Nakamura T, Filho BP, Nakamura CV. Recent advances in leishmaniasis treatment. Int J Infect Dis. 2011 Aug;15(8):e525-32. doi: 10.1016/j.ijid.2011.03.021. Epub 2011 May 24. PMID 21605997
- [Background] Almeida OL, Santos JB. Advances in the treatment of cutaneous leishmaniasis in the new world in the last ten years: a systematic literature review. An Bras Dermatol. 2011 May-Jun;86(3):497-506. doi: 10.1590/s0365-05962011000300012. English, Portuguese. PMID 21738967
- [Background] Silva NS, Muniz VD. [Epidemiology of American tegumentary leishmaniasis in the State of Acre, Brazilian Amazon]. Cad Saude Publica. 2009 Jun;25(6):1325-36. doi: 10.1590/s0102-311x2009000600015. Portuguese. PMID 19503963
- [Background] Soto J, Rea J, Balderrama M, Toledo J, Soto P, Valda L, Berman JD. Efficacy of miltefosine for Bolivian cutaneous leishmaniasis. Am J Trop Med Hyg. 2008 Feb;78(2):210-1. PMID 18256415
- [Background] Blum J, Desjeux P, Schwartz E, Beck B, Hatz C. Treatment of cutaneous leishmaniasis among travellers. J Antimicrob Chemother. 2004 Feb;53(2):158-66. doi: 10.1093/jac/dkh058. Epub 2004 Jan 16. PMID 14729756
- [Background] Blum J, Lockwood DN, Visser L, Harms G, Bailey MS, Caumes E, Clerinx J, van Thiel PP, Morizot G, Hatz C, Buffet P. Local or systemic treatment for New World cutaneous leishmaniasis? Re-evaluating the evidence for the risk of mucosal leishmaniasis. Int Health. 2012 Sep;4(3):153-63. doi: 10.1016/j.inhe.2012.06.004. PMID 24029394
- [Background] Robledo SM, Velez ID, Schmidt TJ. Arnica Tincture Cures Cutaneous Leishmaniasis in Golden Hamsters. Molecules. 2018 Jan 12;23(1):150. doi: 10.3390/molecules23010150. PMID 29329207
- See also: Common Terminology Criteria for Adverse Events (CTCAE) — http://ctep.cancer.gov